CLINICAL TRIAL: NCT06799455
Title: Comparison of Uncuffed Endotracheal Tube to no Endotracheal Tube in EBUS-TBNA Procedure Under Moderate Sedation
Brief Title: Uncuffed Endotracheal Tube vs. no Endotracheal Tube
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACCS-2024-33033
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Multiple Pulmonary Diseases

STUDY DESIGN:
Intervention Model Description: Patient will be randomized 1:1 to UCETT vs no ETT (current standard procedure) when they scheduled for the EBUS-TBNA procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- uncuffed endotracheal group (Experimental)
  Interventions: Device: Endotracheal tube
- no endotracheal tube group/control (No Intervention)

INTERVENTIONS:
Device: Endotracheal tube — participants either receive the ETT during the procedure
  Arms: uncuffed endotracheal group

SUMMARY:
This is a comparison of uncuffed endotracheal tube (UCETT) vs. no endotracheal tube (ETT) in endobronchial ultrasound-transbronchial needle aspiration (EBUS-TBNA) procedure under moderate sedation in terms of procedure tolerance, duration of the procedure, desaturation, amount of sedation medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that is scheduled for EBUS-TBNA procedure

Exclusion Criteria:

* Those who are not safe to receive moderate sedation or flexible bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Desaturation | During the procedure
  Whether a patient will experience any desaturation

CONTACTS AND LOCATIONS:
Overall Officials: H. Erhan Dincer, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States